CLINICAL TRIAL: NCT06110754
Title: Integrative Training Program for Pediatric Sickle Cell Pain (I-STRONG for SCD): Optimizing Feasibility and Acceptability
Brief Title: Development and Adaptation of I-STRONG for SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Soumitri Sil, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005410; R61AT012421-01 (NIH); 2023P005194 (Other: Emory IRB)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell pain; Pediatrics; Mind-body intervention; Behavioral intervention
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Participants in Aim 1 provide feedback for adapting I-STRONG for SCD while participants in Aim 2 receive the I-STRONG for SCD intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Development of I-STRONG for SCD (No Intervention): Adolescents with sickle cell disease and their parents participating completing in-depth interviews over two sessions as part of adapting an integrative, multicomponent, behavioral intervention combining mind-body, cognitive, and behavioral coping skills with neuromuscular exercise training for adolescents with chronic SCD pain.
- I-STRONG for SCD (Experimental): Adolescents with sickle cell disease and their parents participating in a multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training.
  Interventions: Behavioral: I-STRONG for SCD

INTERVENTIONS:
Behavioral: I-STRONG for SCD — I-STRONG for SCD is a group-based, multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training. The intervention includes 16 sessions that occur over 8 weeks. Adolescents attend every session and parents attend 6 of the 16 sessions.
  Arms: I-STRONG for SCD

SUMMARY:
This study develops and tests the feasibility and acceptability of an adapted intervention, Integrative Strong Body and Mind Training (I-STRONG), in adolescents with pain from sickle cell disease.

DETAILED DESCRIPTION:
Pain is the hallmark feature of sickle cell disease (SCD), a life-limiting chronic illness that disproportionately affects African Americans. Well-documented racial disparities complicate effective pain control and the under-treatment of pain experienced by Black Americans with SCD. Approximately 20% of youth with SCD develop chronic pain and experience significant functional impairment, diminished quality of life, and comorbid depression and anxiety that can worsen over time. Youth with chronic SCD pain often are stuck in a vicious cycle of pain, functional impairment, and pain-related fear of movement that contributes to activity avoidance and exacerbates pain. The most effective chronic SCD pain management requires multicomponent, interdisciplinary treatment approaches that include integrative mind-body treatments. Mind-body approaches, specifically diaphragmatic breathing, progressive muscle relaxation, and guided imagery, can improve outcomes for youth with chronic pain. However, multicomponent interventions tailored for chronic SCD pain have never been established. Most pain interventions are developed and studied largely with white youth, do not address cultural influences, and consequently have limited generalizability for minoritized populations that experience health disparities like SCD. There is a critical need for effective, culturally tailored, integrative pain management approaches to address health disparities and improve outcomes for youth with SCD whose chronic pain can persist into adulthood.

To address this unmet need, the researchers will leverage an existing innovative intervention designed for juvenile fibromyalgia, the Fibromyalgia Integrative Training for Teens (FIT Teens). Recent clinical practice guidelines for SCD pain identified fibromyalgia as most closely aligned with chronic pain in SCD to inform treatment recommendations; thus, FIT Teens is well-suited for adaptation and testing for SCD. FIT Teens is an 8-week (16 session) group-based telehealth intervention that combines mind-body, cognitive-behavioral, and neuromuscular movement approaches. Early trials of FIT Teens found excellent patient engagement, and medium to large effects on reducing disability, pain, depressive symptoms, and fear of movement without adverse effects of pain exacerbation. An ongoing multicenter trial of FIT Teens has excellent patient retention (>80%, n=300 enrolled). The mind-body, cognitive-behavioral, and neuromuscular movement treatment components will form the basis of a new multicomponent integrative intervention tailored for SCD.

Aim 1 of this study is to adapt and refine the integrative components of the FIT Teens intervention to develop a new culturally tailored I-STRONG intervention for youth with chronic SCD pain. The investigators will conduct mixed method approaches and purposive sampling to collect qualitative feedback informed by patient and family lived experiences regarding intervention content, format, perceived benefits, and barriers/facilitators to engagement from 15 patients (12 to 18 years of age) with chronic SCD pain and their parents and about 8 adolescents and 8 parents to participate in stakeholder advisory boards. Community stakeholder advisory boards and iterative design will inform intervention adaptation and refinement to enhance clinical implementation. Outcome measures are not collected from participants in Aim 1 as the purpose of this part of the study is to prepare the I-STRONG intervention to be studied for Aim 2.

Aim 2 of the study is to assess feasibility and acceptability of I-STRONG intervention for youth with chronic SCD pain. The investigators will conduct a single-arm proof-of-concept study of the I-STRONG intervention with 12 adolescents (12 to 18 years of age), and the parents of adolescents under the age of 18, to iteratively optimize the feasibility and acceptability of I-STRONG in youth with chronic SCD pain. Feasibility will be demonstrated by rates of study enrollment, retention, and adherence (target goals set at ≥ 75%). Acceptability will be demonstrated by treatment burden, satisfaction, and tolerability. Qualitative feedback about the program format and content will inform additional intervention optimization, refinement, and enhance feasibility and acceptability.

Support from and inclusion in the National Institutes of Health (NIH) Helping to End Addiction Long-term Initiative (HEAL), or NIH HEAL Initiative, is provided for this study. For more information about the initiative visit the HEAL Initiative (https://heal.nih.gov/).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SCD (any genotype)
* Score of at least 3 (indicating medium to high risk for chronic pain) on the Pediatric Pain Screening Tool
* Stable disease-modifying treatments, if applicable, as defined by no newly initiated or significantly increased dosages (mg/kg) in the past 3 months (Aim 2 only)
* English fluency (Aim 2 only)

Exclusion Criteria:

* Comorbid medical conditions typically associated with pain but unrelated to SCD (e.g., rheumatologic disorders or inflammatory bowel disease)
* Presence of a condition(s) or diagnosis, either physical or psychological, or physical exam finding that precludes participation (e.g., severe avascular necrosis with limited or non-weight bearing restrictions, significant cognitive or developmental limitations, active suicidal ideation) (Aim 2 only)
* Adolescent receiving active treatment (e.g., weekly appointments with a provider) for nonpharmacological therapies (e.g, structured behavioral pain management, physical therapy, or acupuncture program) that overlap with the active phase of the study intervention (Aim 2 only)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soumitri Sil, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be available for sharing including study-level metadata and NIH Helping to End Addiction Long-term (HEAL) Common Data Elements.
Time Frame: Data will be available for sharing one year after the end date for this study.
Access Criteria: Data for sharing will be in a public use, NIH HEAL-approved data repository.

REFERENCES:
- [Result] Mooney JT, Sinha C, Bakshi N, Nunez A, Adkins T, Thomas S, Beasley K, Akintobi T, Crosby L, Kashikar-Zuck S, Dampier C, Myer GD, Kesar T, Quinn CT, Sil S. Physical activity among adolescents and young adults living with chronic pain and sickle cell disease: a qualitative examination. J Pediatr Psychol. 2025 Dec 1;50(12):1079-1087. doi: 10.1093/jpepsy/jsaf055. PMID 40694814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta in Atlanta, Georgia, and Cincinnati Children's Hospital Medical Center in Cincinnati, Ohio, USA. Participants for Aim 1 were enrolled June through October 2023. Participant enrollment for Aim 2 began October 24, 2023 and all follow-up assessments were completed by June 14, 2024.
Groups:
- Development of I-STRONG for Sickle Cell Disease (SCD) - Adolescents (Aim 1): Adolescents with sickle cell disease completing in-depth interviews over two sessions as part of adapting an integrative, multicomponent, behavioral intervention combining mind-body, cognitive, and behavioral coping skills with neuromuscular exercise training for adolescents with chronic SCD pain. Outcome measures are not collected from participants in Aim 1 as the purpose of this part of the study is to prepare the I-STRONG intervention to be studied for Aim 2.
- Development of I-STRONG for SCD - Parents (Aim 1): Parents of adolescents with sickle cell disease completing in-depth interviews over two sessions as part of adapting an integrative, multicomponent, behavioral intervention combining mind-body, cognitive, and behavioral coping skills with neuromuscular exercise training for adolescents with chronic SCD pain. Outcome measures are not collected from participants in Aim 1 as the purpose of this part of the study is to prepare the I-STRONG intervention to be studied for Aim 2.
- I-STRONG for Adolescents With SCD (Aim 2): Adolescents with sickle cell disease (SCD) participating in a multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training.
  Integrative Strong Body and Mind Training (I-STRONG) for SCD is a group-based, multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training. The intervention includes 16 sessions that occur over 8 weeks. Adolescents attend each of the 16 sessions.
- I-STRONG for Parents of Adolescents With SCD (Aim 2): Parents of adolescents with sickle cell disease participating in a multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training. Parents are enrolled when the adolescent is under the age of 18.
  I-STRONG for SCD is a group-based, multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training. The intervention includes 16 sessions that occur over 8 weeks. Parents attend 6 of the 16 sessions.
Period: Overall Study
Arm/Group | Development of I-STRONG for Sickle Cell Disease (SCD) - Adolescents (Aim 1) | Development of I-STRONG for SCD - Parents (Aim 1) | I-STRONG for Adolescents With SCD (Aim 2) | I-STRONG for Parents of Adolescents With SCD (Aim 2)
Started | 12 | 12 | 12 | 9
Completed | 12 | 12 | 11 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Development of I-STRONG for SCD - Adolescents (Aim 1): Adolescents with sickle cell disease completing in-depth interviews over two sessions as part of adapting an integrative, multicomponent, behavioral intervention combining mind-body, cognitive, and behavioral coping skills with neuromuscular exercise training for adolescents with chronic SCD pain.
- Development of I-STRONG for SCD - Adults (Aim 1): Parents of adolescents with sickle cell disease completing in-depth interviews over two sessions as part of adapting an integrative, multicomponent, behavioral intervention combining mind-body, cognitive, and behavioral coping skills with neuromuscular exercise training for adolescents with chronic SCD pain.
- I-STRONG for Adolescents With SCD (Aim 2): Adolescents with sickle cell disease participating in the I-STRONG intervention. I-STRONG for SCD is a group-based, multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training. The intervention includes 16 sessions that occur over 8 weeks. Adolescents attend each of the 16 sessions.
- I-STRONG for Parents of Adolescents With SCD (Aim 2): Parents of adolescents with sickle cell disease participating in the I-STRONG intervention. Parents are enrolled when the adolescent is under the age of 18. I-STRONG for SCD is a group-based, multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training. The intervention includes 16 sessions that occur over 8 weeks. Parents attend 6 of the 16 sessions.
- Total: Total of all reporting groups
Arm/Group | Development of I-STRONG for SCD - Adolescents (Aim 1) | Development of I-STRONG for SCD - Adults (Aim 1) | I-STRONG for Adolescents With SCD (Aim 2) | I-STRONG for Parents of Adolescents With SCD (Aim 2) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 9 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 0 | 9 | 0 | 21
  Between 18 and 65 years | 0 | 12 | 3 | 9 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.03 (1.58) | 39.50 (5.63) | 16.30 (1.61) | 40.80 (4.40) | 26.27 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 5 | 9 | 32
  Male | 6 | 0 | 7 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 12 | 8 | 43
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 12 | 12 | 8 | 44
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 12 | 9 | 45
Sickle Cell Disease Genotype [Count of Participants; unit: Participants] — Population: Sickle cell disease genotype is only relevant for adolescent participants with sickle cell disease. Genotypes HbSS and HbSβ0 thalassemia are generally the most severe forms of SCD.
  Participants
    number analyzed (Participants) | 12 | 0 | 12 | 0 | 24
    HbSS (Aim 2) | 0 |  | 8 |  | 8
    HbSC (Aim 2) | 0 |  | 2 |  | 2
    HbSβ+ thalassemia (Aim 2) | 0 |  | 1 |  | 1
    HbSβ0 thalassemia (Aim 2) | 0 |  | 1 |  | 1
    HbSS or HbSβ0 thalassemia (Aim 1 categorization) | 11 |  | 0 |  | 11
    HbSC or HbSβ+ thalassemia (Aim 1 categorization) | 1 |  | 0 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) Pain Severity Score
Description: Pain intensity is rated with the pain severity item of the Brief Pain Inventory (BPI). The single item is scored on a scale from 0 to 10 where no pain = 0 and severe pain = 10.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: The analysis population includes adolescent participants who completed the indicated study visit and completed the survey. One participant withdrew prior to the post-treatment assessment at Week 8 and an additional participant declined to complete the surveys at the 3 months post-treatment assessment at Month 5.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- I-STRONG for Adolescents With Sickle Cell Disease (SCD): Adolescents with sickle cell disease participating in the I-STRONG intervention. I-STRONG for SCD is a group-based, multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training. The intervention includes 16 sessions that occur over 8 weeks. Adolescents attend each of the 16 sessions.
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 12
units on a scale
  Baseline | 5.75 (2.63)
  Post-treatment (Week 8): number analyzed (Participants) | 11
  Post-treatment (Week 8) | 4.36 (1.96)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10
  3 Months Post-treatment (Month 5) | 3.89 (2.15)

2. Secondary Outcome: Brief Pain Inventory (BPI) Pain Interference Score
Description: Functional interference due to pain rated with the impact of pain on daily functions item of the Brief Pain Inventory (BPI). The single item is scored on a scale from 0 to 10 where no pain = 0 and severe pain = 10.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: The analysis population includes adolescent participants who completed the indicated study visit and completed the survey. One participant withdrew prior to the post-treatment assessment at Week 8, an additional participant declined to complete the surveys at the 3 months post-treatment assessment at Month 5, and one participant did not complete this survey during the 3 months post-treatment assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 12
units on a scale
  Baseline | 3.45 (3.09)
  Post-treatment (Week 8): number analyzed (Participants) | 11
  Post-treatment (Week 8) | 4.24 (2.62)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 9
  3 Months Post-treatment (Month 5) | 2.94 (2.15)

3. Secondary Outcome: Patient Health Questionnaire (PHQ-8) Score
Description: Depressive symptoms in past two weeks among adolescent and parent study participants is assessed with the Patient Health Questionnaire (PHQ-8). The PHQ-8 has 8 items that are responded to on a 4-point scale where " not at all" = 0 and "nearly every day" = 3. Total scores range from 0 to 24 where higher scores indicate increased symptoms of depression.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: The analysis population includes adolescent and adult participants who completed the indicated study visit and completed the survey. One adolescent participant withdrew prior to the post-treatment assessment at Week 8 and an additional participant declined to complete the surveys at the 3 months post-treatment assessment at Month 5.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- I-STRONG for Parents of Adolescents With SCD: Parents of adolescents with sickle cell disease participating in the I-STRONG intervention. Parents are enrolled when the adolescent is under the age of 18. I-STRONG for SCD is a group-based, multi-component intervention that includes mind-body, cognitive-behavioral, and neuromuscular movement training. The intervention includes 16 sessions that occur over 8 weeks. Parents attend 6 of the 16 sessions.
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD) | I-STRONG for Parents of Adolescents With SCD
Number analyzed (Participants) | 12 | 9
score on a scale
  Baseline | 6.50 (5.69) | 5.33 (4.8)
  Post-treatment (Week 8): number analyzed (Participants) | 11 | 9
  Post-treatment (Week 8) | 6.82 (6.52) | 5.11 (7.8)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10 | 9
  3 Months Post-treatment (Month 5) | 5.40 (3.41) | 5.22 (7.6)

4. Secondary Outcome: General Anxiety Disorder (GAD-2) Score
Description: General worry in past two weeks among adolescent and parent study participants is assessed with the General Anxiety Disorder (GAD-2) instrument. The GAD-2 has 2 items that are responded to on a 4-point scale where " not at all" = 0 and "nearly every day" = 3. Total scores range from 0 to 6 where higher scores indicate increased experiences of worry.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD) | I-STRONG for Parents of Adolescents With SCD
Number analyzed (Participants) | 12 | 9
score on a scale
  Baseline | 2.08 (1.72) | 2.11 (2.2)
  Post-treatment (Week 8): number analyzed (Participants) | 11 | 9
  Post-treatment (Week 8) | 1.45 (1.44) | 1.11 (1.9)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10 | 9
  3 Months Post-treatment (Month 5) | 1.20 (1.32) | 1.11 (1.9)

5. Secondary Outcome: Pain Catastrophizing Scale Score
Description: Exaggerated worried thoughts of pain are assessed among adolescent and parent study participants. The Pain Catastrophizing Scale, Child and Parent Report, is a 13-item well-validated self-report and parent-report measure of worried thoughts about pain. Items are answered on a 5-point scale where 0 = not true at all and 4 = very true. Total scores range from 0 to 52 and higher scores indicate increased catastrophic thinking.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-Treatment (Month 5)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD) | I-STRONG for Parents of Adolescents With SCD
Number analyzed (Participants) | 12 | 9
score on a scale
  Baseline | 24.33 (13.05) | 28.33 (10.2)
  Post-treatment (Week 8): number analyzed (Participants) | 11 | 9
  Post-treatment (Week 8) | 22.82 (14.06) | 30.56 (9.9)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10 | 9
  3 Months Post-treatment (Month 5) | 21.00 (12.33) | 26.33 (10.7)

6. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL) Score
Description: Health-related quality of life and impact on child and family in the past month is assessed among adolescent study participants with the Pediatric Quality of Life Inventory (PedsQL). The 23-item PedsQL was developed as part of the NIH Roadmap Initiative to create universal measures for patient-reported outcomes and contains questions in the domains of social-peer, depression, anxiety, mobility, and function. Responses are given on a 5-point scale where 0 = never and 4 = almost always. Items are reverse scored and linearly transformed to a scale of 0 to 100, where higher total mean scores indicate a better quality of life.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: The analysis population includes adolescent participants who completed the indicated study visit and completed the survey. One participant withdrew prior to the post-treatment assessment at Week 8 and an additional participant declined to complete the surveys at the 3 months post-treatment assessment at Month 5. This survey was not administered to parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 12
score on a scale
  Baseline | 69.03 (15.03)
  Post-treatment (Week 8): number analyzed (Participants) | 11
  Post-treatment (Week 8) | 64.85 (17.25)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10
  3 Months Post-treatment (Month 5) | 73.83 (16.56)

7. Secondary Outcome: Adolescent Sleep-Wake Scale (ASWS) Score
Description: The Adolescent Sleep Wake Scale (ASWS) is a 28-item patient-reported describing the occurrence and frequency of various behavioral sleep characteristics over the past month. Responses are given on a 6-point Likert scale where 1 = always and 6 = never. Total scores range from 28 to 168 and higher scores indicate better sleep quality.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 12
score on a scale
  Baseline | 38.00 (9.73)
  Post-treatment (Week 8): number analyzed (Participants) | 11
  Post-treatment (Week 8) | 37.55 (9.98)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10
  3 Months Post-treatment (Month 5) | 41.00 (6.58)

8. Secondary Outcome: National Institute on Drug Abuse (NIDA)-Modified ASSIST (NM ASSIST) Tool Level 2
Description: Substance use among adolescent study participants during the past 3 months is assessed with the NIDA-Modified Assist Tool Level 2 for children aged 11-17. The instrument asks respondents how often they have used 15 different substances. Responses are given on a 5-point scale where "not at all" = 0, "less than a day or two" = 1, "several days" = 2, "more than half the days" = 3, and "nearly every day" = 4. Responses to items were then scored as either 0 for non-use of a particular substance or 1 for any use of a particular substance (encompassing scale scores of 1 - 4). The tool is scored as the number of items with a score of greater than 0. The total score ranges from 0 to 15 with higher values indicating use of a greater number of substances.
Time Frame: Baseline, 3 Months Post-treatment (Month 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 12
score on a scale
  Baseline | 0.58 (0.90)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10
  3 Months Post-treatment (Month 5) | 0.50 (0.71)

9. Secondary Outcome: Days of Opioid Use Per Week
Description: Daily use of opioid pain medication is determined based on participant completion of daily diaries for one week at each assessment visit. Participants record opioid use daily as presence or absence of use.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: The analysis population includes participants who completed any number of days of the daily diaries for the indicated time point. Some participants did not complete any diary days.
Measure: Mean (Standard Deviation); unit: days per week of opioid use
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 10
days per week of opioid use
  Baseline: number analyzed (Participants) | 9
  Baseline | 1.00 (2.12)
  Post-treatment (Week 8) | 1.70 (2.49)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 8
  3 Months Post-treatment (Month 5) | 2.25 (2.25)

10. Secondary Outcome: Change in Patient Global Impression of Change (PGIC) Score
Description: The overall self-reported rating of the efficacy of treatment is assessed with the Patient Global Impression of Change (PGIC) instrument. The PGIC asks respondents to rate their overall improvement compared to baseline. Responses are given on a scale of 1 to 7 where 1 = very much improved and 7 = very much worse.
Time Frame: Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: The analysis population includes adolescent participants who completed the indicated study visit and completed the survey. One participant withdrew prior to the post-treatment assessment at Week 8 and two additional participants declined to complete this survey at the 3 months post-treatment assessment at Month 5.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 11
units on a scale
  Baseline to Post-treatment (Week 8) | 1.36 (1.03)
  Baseline to 3 Months Post-treatment (Month 5): number analyzed (Participants) | 9
  Baseline to 3 Months Post-treatment (Month 5) | 1.44 (1.01)

11. Secondary Outcome: Treatment Evaluation Inventory-Short Form (TEI-SF) Score
Description: The Treatment Evaluation Inventory-Short Form is completed at the end of treatment. It includes 9 items adapted to be specific to pediatric pain. Items are rated on a 5-point Likert scale ranging from 1 to 5. Total scores range from 9 to 45. Higher scores indicate increased acceptability with the study treatment.
Time Frame: Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 11
score on a scale
  Post-treatment (Week 8) | 34.36 (4.23)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10
  3 Months Post-treatment (Month 5) | 33.30 (3.23)

12. Secondary Outcome: Tampa Scale of Kinesiophobia (TSK) Score
Description: Fear of movement related to fear of pain is assessed with the Tampa Scale of Kinesiophobia (TSK) instrument. The TSK is a 17-item questionnaire where responses are given on a 4-point Likert scale. Responses of "strongly agree" are coded as 1 and responses of "strongly agree" are coded as 4. Total scores range from 17 to 68 where higher scores indicate greater kinesiophobia.
Time Frame: Baseline, Post-treatment (Week 8), 3 Months Post-treatment (Month 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
Number analyzed (Participants) | 12
score on a scale
  Baseline | 25.42 (6.93)
  Post-treatment (Week 8): number analyzed (Participants) | 11
  Post-treatment (Week 8) | 25.82 (7.24)
  3 Months Post-treatment (Month 5): number analyzed (Participants) | 10
  3 Months Post-treatment (Month 5) | 24.00 (6.78)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from adolescent participants beginning at the baseline assessment and continued through the final assessment at the 3-month post-treatment study visit (up to 5 months).
Description: Adverse events were not collected from parents of adolescent participants. Adverse events were not collected from Aim 1 participants.
Arm/Group | I-STRONG for Adolescents With Sickle Cell Disease (SCD)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I-STRONG for Adolescents With Sickle Cell Disease (SCD) (N=12)
Hospitalization due to pain crisis (General disorders) | 4 (5)
Hospitalization due to body pain and sinus pressure (General disorders) | 1 (1)
Hospitalization due to COVID-19 (Infections and infestations) | 1 (1)
Hospitalization due to pulled muscle with back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I-STRONG for Adolescents With Sickle Cell Disease (SCD) (N=12)
Abdominal pain (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest pain with back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Mild bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness in lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (2)
Pain crisis (General disorders) | 1 (1)
Passive suicidal ideation (Psychiatric disorders) | 1 (1)
Sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Stress (Social circumstances) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT06110754/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT06110754/ICF_000.pdf